CLINICAL TRIAL: NCT02253563
Title: Resistance Training Versus Balance Training to Improve Postural Control in Patients With Parkinson's Disease - a Randomized Controlled Rater Blinded Trial
Brief Title: Resistance Versus Balance Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Christian Schlenstedt, PhD, University of Kiel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A 146/11
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance Training (Experimental): Group performing resistance training.
  Interventions: Behavioral: Resistance Training
- Balance Training (Experimental): Group performing balance training.
  Interventions: Behavioral: Balance Training

INTERVENTIONS:
Behavioral: Resistance Training
  Arms: Resistance Training
Behavioral: Balance Training
  Arms: Balance Training

SUMMARY:
Comparison of resistance training versus balance training to improve postural control in patients with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's Disease, postural instable

Exclusion Criteria:

* cardiopulmonary/metabolic diseases that could interfere with the safe conduct of the study protocol, unstable medication, severe cognitive impairments that do not allow the patients to follow exercise instructions, participation in a resistance or balance training program (beside usual physical therapy), Deep Brain Stimulation.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Fullerton Advanced Balance scale | up to 2 years

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Schlenstedt C, Paschen S, Kruse A, Raethjen J, Weisser B, Deuschl G. Resistance versus Balance Training to Improve Postural Control in Parkinson's Disease: A Randomized Rater Blinded Controlled Study. PLoS One. 2015 Oct 26;10(10):e0140584. doi: 10.1371/journal.pone.0140584. eCollection 2015. PMID 26501562